CLINICAL TRIAL: NCT02465476
Title: Rationalization of the Treatment Pathway of Patient Suffering From Rare Skin Disease With Telemedicine
Acronym: Telemalrares
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/13/6901
Record Dates: First submitted 2015-04-24; First posted 2015-06-08 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Skin Disease
Keywords: skin disease; telemedicine
MeSH Terms: conditions — Skin Diseases | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal care (No Intervention): patient who will have normal treatment pathway
- telemedicine (Experimental): patient who will have telemedicine
  Interventions: Procedure: telemedicine

INTERVENTIONS:
Procedure: telemedicine — treatment pathway organized by telemedicine
  Arms: telemedicine

SUMMARY:
The investigators want to demonstrate that a new organization with telemedicine could rationalize the treatment pathway of patient suffering from rare skin disease. A diagnosis and a personalised treatment pathway could be performed before the consultation in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* New patients suffering from a rare skin disease whatever pathology or age, which needs a take-over by this centre
* Or patients already take-over by the centre but lost to follow-up for more than one year
* Patients (and/or parents) who give their consents
* Patients (and/or parents) able to fill in questionnaires

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Patients subject to a judicial safeguard order
* Patients who need an emergency take-over
* Patients followed by a doctor who does not have a computerized system or refuse to send data via the secured messaging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Number of hospital visits | 6 months
  Interest of a procedure of telemedicine on the organization of the treatment pathway of patients affected by rare skin diseases in terms of change of the number of visit in hospital.

SECONDARY OUTCOMES:
Improvement of the treatment pathway and its organization | 6 months
  Traceability in the information system by composite criteria : number of completed application forms, number of meeting per month, number of meeting a month, number of patients treated a month, time dedicated to the logistical coordination (collection by sheets of weekly time) and number of new patients per month.
Satisfaction of the patient | 6 months
  questionnaire of satisfaction Short Form-36 Health Survey (SF36)
Change of the cost related to the patient care (direct and indirect). | 6 months
  Composite criteria with number of consultations and hospitalizations, number of visit in hospital and number of days of work and school absenteeism.
management of time by the medical personal. | 6 months
  collection by sheets of weekly time

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Mazereeuw-Hautier, MD . PHD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France